CLINICAL TRIAL: NCT05677139
Title: Asthma Control in Severe Asthma Patients Treated With Tezepelumab: A Prospective, Observational, Real-World Evidence Study (ASCENT)
Brief Title: A Study for Observing Severe Asthma in Patients Treated With Tezepelumab
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5180R00011
Record Dates: First submitted 2022-11-29; First posted 2023-01-10 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Asthma
Keywords: Real-World Evidence; Severe Uncontrolled Asthma; Inhaled corticosteroids (ICS); Post-Authorization
MeSH Terms: conditions — Asthma | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective Cohort: Participants with severe uncontrolled asthma will receive tezepelumab. Relevant demographics, baseline clinical data, and asthma control questionnaire-6 (ACQ-6) will be retrospectively collected. All patient reported outcomes (PROs) will be prospectively collected. Other outcomes of interest (tezepelumab patterns of utilization, lung function, asthma exacerbations, medication use, and healthcare resource utilization [HRU]) will be collected at baseline (retrospective collection for 52-week pre-index period during enrolment) and prospectively collected during enrolment for participants who enroll into the study before the first dose of tezepelumab, and for a period of up to 52 weeks (at Weeks 4, 12, 24, and 52) after the index date. The index date is defined as the date when participants receive the first dose of tezepelumab.
  Interventions: Other: None (Observational Study)

INTERVENTIONS:
Other: None (Observational Study) — Not applicable since it's an observational study.
  Other Names: Observational Study

SUMMARY:
A study involving primary data collection within real-world settings of participants who initiate treatment with tezepelumab for severe uncontrolled asthma. This study will complement evidence obtained from randomized controlled trials and provide new data focusing on the holistic and patient reported outcome (PRO).

DETAILED DESCRIPTION:
This is a 12-month, multi-country, multi-center, prospective, non-comparative and non-interventional (observational), post-reimbursement real-world evidence study that will assess asthma symptom control, lung function, and patient-reported outcomes including health-related quality of life after tezepelumab treatment initiation in participants with severe asthma in Europe and Canada. This study is planned to be conducted in several countries including but not limited to Canada, Germany, Denmark, Switzerland, and Sweden.

Participants will be followed for a maximum period of 52 weeks after tezepelumab treatment initiation, irrespective of treatment discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged 12 years or older
* Provision of signed and dated written informed consent, including assent for minors
* Prescribed treatment with Tezepelumab
* Diagnosis of asthma for at least 52 weeks prior to enrolment date and symptoms confirmed by the Investigator not to be due to alternative diagnoses
* Received at least one prescription of medium-dose to high-dose inhaled corticosteroids (ICS) during the 52 weeks prior to enrolment date
* Use of additional asthma maintenance controller medication(s) for at least 52 weeks prior to enrolment date
* Documented history of at least 1 asthma exacerbations during the 52 weeks prior to enrolment date
* Individuals with ACQ-6 score ≥ 1.5 (indicating inadequate asthma symptom control) at enrolment or up to 12 weeks before enrolment
* Participants currently receiving care from pulmonologists and/or allergists
* Participants who are able to understand and complete the ePROs
* Availability of participants medical records for asthma exacerbation and Healthcare Resource Utilization (HCRU) for the 52 weeks prior to Tezepelumab initiation

Exclusion Criteria:

* Any contraindication to Tezepelumab
* Participants on concurrent biologics for asthma at the time of receiving the first dose of Tezepelumab will be excluded except for stable allergen immunotherapy (defined as a stable dose and regimen at the time of enrolment)
* Participation in an observational study that might, in the Investigator's opinion, influence the assessment for the current study, or participation in an interventional clinical trial in the last 3 months
* Pregnancy or lactation period.

Ages: 12 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants aged 12 years or older with severe uncontrolled asthma who will commence treatment with Tezepelumab and will be enrolled from a diverse population of clinical settings. In the first wave, the study population is planned to comprise approximately 200 participants with an additional 200 participants in the second wave.
Sampling Method: Non-Probability Sample
Enrollment: 513 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Asthma Control Questionnaire (ACQ-6) score | Week 52
  Participant-reported asthma symptom control using ACQ-6 will be described. The ACQ-6 was developed for self-administration by adults and adolescents by omitting the forced expiration volume in 1 second (FEV1) % predicted question. Patients are asked to record their experience with 5 symptoms (night-time waking, symptoms on waking, activity limitation, shortness of breath, and wheezing) and use of short-acting. β2 agonist over the previous week using a 7-point scale (0 = no impairment; 6 = maximum impairment). The ACQ-6 score is calculated by taking the mean of the 6 equally weighted items. The ACQ-6 score range is 0 (well controlled) to 6 (extremely poorly controlled).
Change in Asthma Control Questionnaire 6 (ACQ-6) score from Baseline | From Baseline (Week -52 to Week 0) to Week 52
  Participant-reported asthma symptom control using ACQ-6 will be described. The minimum value of ACQ-6 score is 0 and the maximum value of ACQ-6 score is 6. The ACQ-6 score of 0 indicates well tolerated asthma whereas, the ACQ-6 score of 6 indicates extremely poorly controlled asthma
Number of participants with improvement in ACQ-6 response score | From Baseline (Week -52 to Week 0) to Week 52
  Improvement from baseline in ACQ-6 score of >=0.5 will be described.
Number of participants with well-controlled asthma (ACQ-6 score ≤ 0.75) | Week 52
  Participant-reported asthma symptom control using ACQ-6 will be described.
Time to first ACQ-6 response | From Baseline (Week -52 to Week 0) to Week 52
  Time to first ACQ-6 response will be assessed. The ACQ-6 response is defined as change from baseline in ACQ-6 score <= -0.5.

SECONDARY OUTCOMES:
St. George's Respiratory Questionnaire (SGRQ) total score | Week 52
  Asthma-specific health-related quality of life (HRQoL) will be described. The SGRQ is a 50-item PRO instrument developed to measure the health status of patients with airway obstruction diseases. The total score indicates the impact of disease on overall health status. This total score is expressed as a percentage of overall impairment, in which 100 represents the worst possible health status and 0 indicates the best possible health status.
Asthma Control Test (ACT) total score | Week 52
  Asthma-specific HRQoL will be described. The ACT is a questionnaire that assesses shortness of breath and general asthma symptoms, use of rescue medications, effect of asthma on daily functioning, and overall asthma control. Patients are asked to recall how their asthma has been during the past 4 weeks by responding to 5 questions on a scale of 1 to 5. The responses from the 5 items are summed to produce an ACT score that range from 5 (poorly controlled asthma) to 25 (well-controlled asthma). An ACT score ≥ 20 indicates well-controlled asthma, 16 to 19 indicates not well-controlled asthma, and ≤ 15 indicates very poorly controlled asthma.
Change from baseline in SGRQ total score | From Baseline (Week -52 to Week 0) to Week 52
  Asthma-specific HRQoL will be described.
Change from baseline in ACT total score | From Baseline (Week -52 to Week 0) to Week 52
  Asthma-specific HRQoL will be described.
Number of participants with improvement in SGRQ total score | From Baseline (Week -52 to Week 0) to Week 52
  Improvement of ≥ 4 in SGRQ total score will be described.
Number of participants with improvement in ACT total score | From Baseline (Week -52 to Week 0) to Week 52
  Improvement of ≥ 3 in ACT total score will be described.
Pre-bronchodilator forced expiratory volume in 1 second (FEV1) | Week 52
  Lung function will be described.
Post-bronchodilator (BD) forced expiratory volume in 1 second (FEV1) | Week 52
  Lung function will be described.
Pre BD forced vital capacity (FVC) | Week 52
  Lung function will be described.
Post-BD FVC | Week 52
  Lung function will be described.
Pre-BD forced expiratory flow (FEF) | Baseline (Week -52 to Week 0), Week 4, Week 24, and Week 52
  Lung function will be described.
Changes from baseline in pre-BD FEF | From Baseline (Week -52 to Week 0) to Week 52
  Lung function will be described.
Changes from baseline in pre-BD FEV1 | From Baseline (Week -52 to Week 0) to Week 52
  Lung function will be described.
Changes from baseline in post-BD FEV1 | From Baseline (Week -52 to Week 0) to Week 52
  Lung function will be described.
Changes from baseline in pre-BD FVC | From Baseline (Week -52 to Week 0) to Week 52
  Lung function will be described.
Changes from baseline in post-BD FVC | From Baseline (Week -52 to Week 0) to Week 52
  Lung function will be described
Proportion of participants with spirometry and/or body plethysmography parameters | Week 52
  Participants will be assessed through spirometry and body plethysmography parameters
Number of participants who achieve 5% or 100 mL improvement in pre-BD and post-BD FEV1 | From Baseline (Week -52 to Week 0) to Week 52
  Lung function will be described.
Annualized asthma exacerbation rate (AAER) | From Baseline (Week -52 to Week 0) to Week 52
  Annual asthma exacerbation rate is calculated in years as total number of exacerbations of interest divided by the total time at risk.
Proportion of participants with asthma exacerbations | From Baseline (Week -52 to Week 0) to Week 52
  Asthma exacerbations will be described.
Proportion of participants with reduced total number of asthma exacerbations | From Baseline (Week -52 to Week 0) to Week 52
  Proportion of participants with reduced total number of asthma exacerbations at the end of 52 weeks compared with baseline
Proportion of participants who completed 52 weeks of tezepelumab treatment with at least 50% reduction in exacerbations | From Baseline (Week -52 to Week 0) to Week 52
  Asthma exacerbations will be described.
Proportion of participants who completed 52 weeks of tezepelumab treatment without an asthma exacerbation | From Baseline (Week -52 to Week 0) to Week 52
  Asthma exacerbations in 52 weeks will be described.
Change from baseline in AAER | Baseline (Week -52 to Week 0) to Week 52
  Asthma exacerbations will be described.
Cumulative asthma exacerbation days | From Baseline (Week -52 to Week 0) to Week 52
  Asthma exacerbations in participants resulting in any hospitalization will be described.
Proportion of participants with any systemic corticosteroid (SCS) or inhaled corticosteroid (ICS) use | From Baseline (Week -52 to Week 0) to Week 52
  Asthma related SCS or ICS use will be described.
Number of participants with categorised percent reduction on cumulative systemic corticosteroids (SCS) dose | From Baseline (Week -52 to Week 0) to Week 52
  Percent reduction on cumulative SCS dose is categorized as follows: >=25%, >=50%, >75% and 100%.
Median SCS or ICS dose change | From Baseline (Week -52 to Week 0) to Week 52
  Asthma related SCS or ICS use will be described.
Proportion of participants with long-term SCS and ICS use | From Baseline (Week -52 to Week 0) to Week 52
  Asthma related SCS or ICS use (>30 consecutive days) before and after tezepelumab initiation will be described.
Time to earliest use SCS from tezepelumab initiation among patients that used SCS or ICS | From Baseline (Week -52 to Week 0) to Week 52
  Time to earliest use SCS from tezepelumab initiation among patients that used SCS or ICS will be described.
Number and type of asthma related healthcare resource utilization (HCRU) | Baseline (Week -52 to Week 0), Week 4, Week 12, Week 24, and Week 52
  Asthma related HCRU will be described.
Annualized rates of asthma-related visits leading to hospitalization and emergency department (ED) visits, urgent care visits, or unscheduled out-patient or physician visits | Baseline (Week -52 to Week 0), Week 4, Week 12, Week 24, and Week 52
  Asthma related HCRU will be described.
Annualized rates of asthma related physician/healthcare calls/visits | From Baseline (Week -52 to Week 0) to Week 52
  Asthma related HCRU will be described.
Duration of asthma-related hospitalisation | From Baseline (Week -52 to Week 0) to Week 52
  Asthma related HCRU will be described.
Proportion of participants with stable disease | From Baseline (Week -52 to Week 0) to Week 52
  Asthma disease stability is a composite endpoint consisting of ACQ-6, FEV1, exacerbations, and OCS use. The participants achieve full disease stability when they reach a meaningful improvement in all 4 parameters which is maintained to the end of the follow-up period (Week 52). This includes ACQ-6 < 1.5, Pre-BD FEV1 at Week 52/pre-BD FEV1 at baseline >0.95, 50% reduction in annualized number of exacerbations in the follow-up period, and at least ≥50% reduction in OCS use in the follow-up period.
Duration (days) of tezepelumab treatment | From Baseline (Week -52 to Week 0) to Week 52
  Tezepelumab treatment features, including duration of therapy will be described.
Proportion of participants with tezepelumab discontinuation and reason(s) | From Baseline (Week -52 to Week 0) to Week 52
  Tezepelumab treatment features, including discontinuation and reasons for discontinuation will be described.
Proportion of participants with switching to other biologics for asthma and reasons(s) | From Baseline (Week -52 to Week 0) to Week 52
  Tezepelumab discontinuation and reasons for discontinuation will be described.
Time to tezepelumab discontinuation | From Baseline (Week -52 to Week 0) to Week 52
  Time taken to discontinue tezepelumab will be described.

CONTACTS AND LOCATIONS:
Locations (60):
- Austria (3):
  - Research Site, Innsbruck
  - Research Site, Klagenfurt Am W Rthersee
  - Research Site, Vienna
- Belgium (6):
  - Research Site, Erpent
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Mouscron
  - Research Site, Woluwe-Saint-Lambert
  - Research Site, Yvoir
- Canada (8):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Colombia
  - Research Site, Kingston, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Montr Al,, Qu Bec
  - Research Site, Saskatoon, Saskatchewan
- Denmark (3):
  - Research Site, Copenhagen
  - Research Site, Hvidovre
  - Research Site, Vejle
- Germany (20):
  - Research Site, Aschaffenburg
  - Research Site, Auerbach
  - Research Site, Augsburg
  - Research Site, Bamberg
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Cottbus
  - Research Site, Düsseldorf
  - Research Site, Flensburg
  - Research Site, Freiburg im Breisgau
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Leipzig
  - Research Site, Marburg
  - Research Site, München
  - Research Site, Schleswig
  - Research Site, Stuttgart
  - Research Site, V Lklingen
  - Research Site, Wiesbaden
- Israel (3):
  - Research Site, Jerusalem
  - Research Site, Rehovot
  - Research Site, Tel Aviv
- Italy (11):
  - Research Site, Ancona
  - Research Site, Bergamo
  - Research Site, Catanzaro
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Palermo
  - Research Site, Roma
  - Research Site, Siena
  - Research Site, Yradate
- Sweden (2):
  - Research Site, Stockholm
  - Research Site, Uppsala
- Switzerland (4):
  - Research Site, Basel
  - Research Site, Chur
  - Research Site, Lugano
  - Research Site, Sion

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from
  AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home